CLINICAL TRIAL: NCT06901583
Title: Impact of a Mindfulness-Oriented Psychoeducational Program on the Mindfulness, Anger and Interpersonal Relationship Styles of Nursing Students: A Randomized Controlled Trial
Brief Title: Impact of a Mindfulness-Oriented Psychoeducational Program on the Mindfulness, Anger and Interpersonal Relationship Styles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Eda Mert, Dr. Eda Mert, Principle Investigator, Aydin Adnan Menderes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/019; HF-22004 (Other Grant/Funding Number: Scientific Research Projects Unit of Aydın Adnan Menderes University)
Record Dates: First submitted 2025-03-21; First posted 2025-03-30 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Nurse's Role; Anger; Interpersonal Relations
Keywords: Mindfulness; Anger; Anger expression; Interpersonal relationship style; Nursing students; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-oriented psychoeducational program (Experimental): The program, consisting of six sessions and developed by evaluating studies in the literature, covers topics such as mindfulness, anger, and interpersonal relationships
  Interventions: Other: Mindfulness-oriented psycho-education

INTERVENTIONS:
Other: Mindfulness-oriented psycho-education — The program, consisting of six sessions and developed by evaluating studies in the literature, covers topics such as mindfulness, anger, and interpersonal relationships

SUMMARY:
Aim: This study aimed to investigate the impact of a mindfulness-oriented psychoeducational program on nursing students' levels of mindfulness, anger, anger expression, and interpersonal relationship styles.

Background: Mindfulness of anger, which significantly influences interpersonal relationships, is especially crucial for the professional practice of nursing. Although numerous studies have explored anger and interpersonal relationships among nursing students, research on the impact of mindfulness interventions within this context remains limited.

Design: This study was a single-blind, randomized controlled trial with pre-test, post-test, and one-month and three-month follow-up assessments.

Methods: The study was conducted at the Faculty of Nursing, Aydın Adnan Menderes University, during the 2022-2023 academic year with first-year nursing students. A total of 84 students (Experimental: 42, Control: 42) were included in the study sample, determined through randomization. The experimental group participated in a six-week mindfulness-oriented psychoeducational program, with weekly sessions lasting 60 to 90 minutes. Data were collected using the Personal Information Form, the Mindful Attention Awareness Scale (MAAS), the Trait Anger/Anger Expression Inventory (TAXI), and the Interpersonal Style Scale (ISS).

ELIGIBILITY:
Inclusion Criteria:

* To have higher mean scores of "trait anger"

Exclusion Criteria:

* Completion of formal training in mindfulness, anger, and interpersonal relationships

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
(MAAS) Mindful Attention Awareness Scale | 3 months
  Effective results-higher scores indicate greater mindfulness
(TAXI) Trait Anger/Anger Expression Inventory | 3 months
  Effective results-higher scores of trait anger, anger-in, and anger-out indicate negative anger; higher scores of anger control indicate greater anger control ability
(ISS) Interpersonal Styles Scale | 3 months
  Non-effective results-higher scores indicate negative interpersonal styles

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Nursing Faculty, Aydin, Turkey (Türkiye)